CLINICAL TRIAL: NCT06189963
Title: A Phase I/IIa, Study to Evaluate the Safety, Tolerability and Exploratory Efficacy of SNK01 in Participants With Moderate Alzheimer's Disease
Brief Title: Clinical Study of SNK01 in Participants With Moderate Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NKGen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNK01-AD01
Record Dates: First submitted 2023-12-06; First posted 2024-01-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Moderate Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SNK01 (Experimental): SNK01 will be administered as an IV infusion Q3W for up to 1 year.
  Interventions: Biological: SNK01
- Placebo (Placebo Comparator): Placebo will be administered as an IV infusion Q3W for up to 1 year.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SNK01 — SNK01 is a novel cell-based, patient specific ex vivo expanded autologous natural killer (NK) cell, immunotherapeutic drug
  Arms: SNK01
Other: Placebo — Sodium Lactate Hartmann's Solution
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test SNK01 in participants with moderate Alzheimer's Disease. The main questions it aims to answer are:

1. Is SNK01 safe and tolerable when administered every 3 weeks for up to 1 year as an intravenous infusion
2. Can SNK01 administration improve cognitive assessment scores and biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. The participant or their legally authorized representative must be willing and able to give their informed consent in writing and comply with the requirements of this study protocol. Informed consent for participants or their legally authorized representative and caregivers will be obtained before any trial-related activity. (Trial-related activities are any procedure that would not be performed during normal treatment of the participant).
2. Participants must have a reliable study partner/caregiver (per investigator judgement for instance a family member, partner etc., guardian (must be always the same person)) who is in close contact with the patient, available on call and who is able to contribute to the assessment of the ratings of the functional endpoints at specific study visits. This person will be able to communicate in the language in which the participant is being assessed and should also serve as a backup contact for the study site. The study partner/caregiver must sign a separate informed consent form which describes their contributions during the study.
3. Patients with diagnosis of Alzheimer's dementia according to the recommendations from the 2011 National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease.
4. Age 40 to 85 years old.
5. Patients must have at least 6 years of formal education and fluency in the test language as verbally confirmed by the patient or their legally authorized representative and documented by the study investigator.
6. Female participants of childbearing potential must have a negative urine pregnancy test at Screening and Visit 1 before first administration of the study drug. Females of childbearing potential are defined as those who are not surgically sterile or who are not post-menopausal (i.e.: no menses for at least 1 year). Male and female participants of reproductive potential must also agree to abstinence or use acceptable form(s) of effective contraception during the study and for 30 days after the final dose of the study drug. Acceptable methods of contraception include the following:

   1. Condoms, sponges, foams, gels, diaphragms, or intrauterine device (IUD).
   2. Hormonal birth control for 30 days prior to administration of the study drug.
   3. A vasectomized sexual partner.
7. Positive evidence for a diagnosis of AD via amyloid positron emission tomography (Amyloid PET) of the brain within the past six months.
8. CDR-SB score of ≥ 9.5 and <16.0.

Exclusion Criteria:

1. Substantial concomitant cerebrovascular disease defined as Fazekas Grade 3.
2. History of a stroke/intracranial hemorrhage temporally related to the onset of worsening of cognitive impairment in the opinion of the investigator.
3. Any substance use disorder that has not been in remission for at least 12 months
4. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.
5. Uncontrolled cardiovascular illnesses such as chronic congestive heart failure (with or without oedema), tachycardia, arrhythmias, uncontrolled hypertension.
6. History of cerebrovascular accident or transient ischemic attack (TIA), or unexplainable loss of consciousness within the last year.
7. Significant pulmonary disease predisposing to hypoxia.
8. Significant ischemic heart disease, myocardial infarction within the last two years and/or with residual angina, orthopnea, conduction defects (ECG), or any other clinically significant heart disease classified as NYHA III or IV.
9. Significant liver disease (for example cirrhosis, active hepatitis B and C, primary or metastatic liver neoplasm).
10. Indication of liver disease, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined during screening.
11. Significant gastrointestinal disorders (for example gastrointestinal bleeding within the last two years, malabsorption syndromes, post-gastrectomy, or active peptic ulcer disease).
12. Immunological disorder such as per investigator judgement clinically significant allergies, Lupus erythematodes, or scleroderma.
13. Uncontrolled/Unstable hematological disease (regardless of cause) such as refractory anemia or refractory myelosuppression.
14. Neurological disease (such as: Lewy body dementia - primary diagnosis, Huntington's disease, Parkinson's Disease, encephalitis, epilepsy, vascular or multi-infarct dementia, stroke, congenital mental deficiency, multiple sclerosis) and psychiatric disorders (such as schizophrenia, or intellectual disability), or any other disorders impacting cognitive function.
15. Unstable/uncontrolled major depression or anxiety within the last 12 months.
16. History of seizures in the past three years.
17. Uncontrolled endocrine disease such as uncontrolled diabetes mellitus or manifest hyperthyroidism, in the opinion of the investigator.
18. Severe renal impairment defined as a GFR < 30 mL/min/1.73 m2 in the screening lab report
19. Infection with human immunodeficiency virus (HIV), hepatitis B, hepatitis C, or any other infection or active systemic disease.
20. Currently being treated with anticoagulants (except aspirin at or below a prophylactic dose).
21. Participants who are taking medications for AD, like memantine or acetylcholinesterase inhibitors (AChEI) that exceeds the normal recommended dose range or have not achieved a stable dose for the 30 days prior to enrollment.
22. Any contraindication for performing a brain MRI and/or Amyloid PET scan.
23. Any participant whose safety the investigator considers to be at risk from this trial's intervention.
24. Participants with any medically unstable/uncontrolled conditions.
25. Any suicidal behavior in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
26. Any suicidal ideation of type 4 or 5 in the C-SSRS in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicity | 3 weeks
  DLTs will be assessed by the review of labs, PE and AEs
Maximum tolerated dose determination | 3 weeks
  Determine the maximum tolerated dose based on the evaluation of the number of participants who experience a DLT which will then determine the RP2D.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 1 Year
  Evaluate the safety and tolerability of SNK01 assessed by labs, PE and AEs
Preliminary efficacy in cognitive assessment scores of CDR-SB | 1 Year
  Measure changes in cognitive assessment of CDR-SB from baseline
Preliminary efficacy in cognitive assessment scores of MMSE | 1 Year
  Measure changes in cognitive assessment of MMSE from baseline
Preliminary efficacy in cognitive assessment scores of NPI | 1 Year
  Measure changes in cognitive assessment of NPI from baseline
Preliminary efficacy in cognitive assessment scores of ADCS-ADL-Severe | 1 Year
  Measure changes in cognitive assessment of ADCS-ADL-Severe from baseline
Preliminary efficacy in cognitive assessment scores of ADAS-Cog | 1 Year
  Measure changes in cognitive assessment of ADAS-Cog from baseline

SECONDARY OUTCOMES:
Changes in CSF biomarkers (pTau 181, Aβ42/40, GFAP, NfL) | 1 Year
  Measure changes in CSF biomarkers as changed from baseline
Changes in plasma biomarkers (pTau 181, Aβ42/40, GFAP, NfL) | 1 Year
  Measure changes in Plasma biomarkers as changed from baseline

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Behavioral Research Specialists, LLC, Glendale, California
  - Syrentis Clinical Research, Santa Ana, California
  - Valiance Clinical Research, Tarzana, California
  - AdventHealth Research Institute, Orlando, Florida
- Ottawa Memory Clinic, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No